CLINICAL TRIAL: NCT02968550
Title: Shunt Evaluation With ALPE System in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, MD, Università degli Studi di Ferrara
Other Study IDs: SEAT
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Mechanical Ventilation; Thoracic Diseases
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low shunt group: patients with shunt less than 30% in one-lung ventilation at ZEEP
- High shunt group: Patients with shunt equal or more than 30% in one-lung ventilation at ZEEP

SUMMARY:
. The aim of this study, thus, is to evaluate shunt fraction and markers of alveolar distress during one lung ventilation (OLV) at different levels of positive end expiratory pressure (PEEP). Moreover, investigators will focus on predicting factors of high shunt levels during OLV.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for thoracoscopic lobectomy or thoracoscopic wedge resection in lateral decubitus.
* patients American Society of Anesthesiologists Physical Status Classiﬁcation score of 1-3

Exclusion Criteria:

* Patients with hemodynamic instability,
* Patients with severe chronic respiratory failure
* Patients with preoperative anemia (hemoglobin <10 g 100 ml-1)
* Patients requiring unplanned conversion to thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracoscopic surgery
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary shunt evaluated with ALPE system | every 30 minutes after the start of surgery up to 3 evaluations, up to 90 minutes

SECONDARY OUTCOMES:
predictors of high intraoperative shunt | The outcome is assessed 15 minutes after one lung ventilation
  All patients admitted to the study received a preoperative physiologic assessment with a cardiovascular evaluation and spirometry. After 15 minutes of one lung ventilation, the pulmonary shunt is evaluated. Therefore, all clinical variable evaluated during preoperative assessment will be compared with the pulmonary shunt

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy

REFERENCES:
- [Background] Beck DH, Doepfmer UR, Sinemus C, Bloch A, Schenk MR, Kox WJ. Effects of sevoflurane and propofol on pulmonary shunt fraction during one-lung ventilation for thoracic surgery. Br J Anaesth. 2001 Jan;86(1):38-43. doi: 10.1093/bja/86.1.38. PMID 11575407